CLINICAL TRIAL: NCT03113253
Title: The Effect of Tranexamic Acid (TXA) on Blood Loss in Burn Surgery - A Randomized, Double-Blinded Placebo-Controlled Trial
Brief Title: TRANexamic Acid to Reduce Bleeding in BURN Surgery
Acronym: TRANBURN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Collaborators: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRANBURN
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Tranexamic Acid; Burns; Surgery; Wounds and Injuries
Keywords: Tranexamic Acid; Burn; Surgery; Excision
MeSH Terms: conditions — Burns; Wounds and Injuries | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Experimental): Patient will receive:
  * 1g of tranexamic acid by slow intravenous injection
  * 1g of tranexamic acid by syringe pump during 8 hours
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Patient will receive:
  * 10 mL of 0.9% sodium chloride by slow intravenous injection
  * 48 mL of 0.9% sodium chloride by syringe pump during 8 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid
  Other Names: Exacyl
  Arms: Tranexamic Acid
Drug: Placebo — 0.9% sodium chloride to mimic tranexamic acid
  Other Names: 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
Excision and grafting in burn patients can lead to severe blood loss. A preliminary study conducted in Saint Joseph Saint Luc Hospital showed that the total median blood loss was 1412 mL (1). Transfused patients had a total median blood loss of 2468 mL and an average number of 4 packed red blood cells (PRBC) administered.

Among the various methods that help limit blood loss, tranexamic acid, which has been proved useful in traumatology and surgery, has not been sufficiently studied in burn patients. A preliminary study in 27 burned patients showed a reduction of blood loss with tranexamic acid (2).

Objective of TRANBURN study is to demonstrate that tranexamic acid help limit blood loss and reduces the use of blood products.

DETAILED DESCRIPTION:
The first aim of the study is to demonstrate that tranexamic acid help limit blood loss and reduces the use of blood products.

Secondary objectives are to evaluate impact of tranexamic acid on mortality, success of skin grafts and occurrence of deep vein thrombosis or myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing burn excision surgery for standard of care purposes
* Male or female >= 18 years of age
* Subject or subject's medical decision maker agrees to participate in this study and provides informed consent

Exclusion Criteria:

* Subjects with a history of hypercoagulopathy, deep vein thrombosis (DVT), pulmonary embolism
* Renal impairment
* Subjects with known hypersensitivity to tranexamic acid
* Consecutive fibrinolytic states to coagulopathy
* History of convulsions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Blood loss (mL / cm² excised) | Until day 5 post surgery
  To determine the impact of tranexamic acid on blood loss in burn surgeries

SECONDARY OUTCOMES:
Need for transfusion | Until day 5 post surgery
  Number of blood product transfused
All-cause Hospital Mortality | Until day 15 post surgery
  Any death during hospital stay
Success of skin graft | Until day 15 post surgery
  Number of successful skin graft (medical assessment)
Deep vein thrombosis | Until day 15 post surgery
  Number of deep vein thrombosis
Myocardial infarction | Until day 15 post surgery
  Number of myocardial infarctions
Stroke | Until day 15 post surgery
  Number of strokes
Pulmonary embolism | Until day 15 post surgery
  Number of pulmonary embolisms
Convulsion | Until day 15 post surgery
  Number of convulsions

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Fontaine, MD, PhD, Principal Investigator — Saint Joseph Saint Luc Hospital, Burn Intensive Care Unit
Locations (4):
- France (4):
  - Service de réanimation des brûlés de Mercy (CHR Metz-Thionville), Ars-Laquenexy
  - Centre Commun de Traitement des Brûlés - Hôpital Edouard Herriot, Lyon
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Centre des brûlés inter-régional Méditerranée - Hôpital de la Conception, Marseille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farny B, Fontaine M, Payre J, Ravat F, Poupelin J-C, Latarjet J. Évaluation des pertes sanguines lors des chirurgies d'excision-autogreffe de peau chez les patients brûlés. Anesthésie & Réanimation. 2015;1:A307-8.
- [Background] Jennes S, Degrave E, Despiegeleer X, Grenez O. Effect of Tranexamic Acid on Blood Loss in Burn Surgery: A Preliminary Study. Journal of Burn Care & Rehabilitation. 2003;24:S59.
- [Background] Mercuriali F, Inghilleri G. Proposal of an algorithm to help the choice of the best transfusion strategy. Curr Med Res Opin. 1996;13(8):465-78. doi: 10.1185/03007999609115227. PMID 9010613
- [Background] Ker K, Edwards P, Perel P, Shakur H, Roberts I. Effect of tranexamic acid on surgical bleeding: systematic review and cumulative meta-analysis. BMJ. 2012 May 17;344:e3054. doi: 10.1136/bmj.e3054. PMID 22611164
- [Background] Zufferey P, Merquiol F, Laporte S, Decousus H, Mismetti P, Auboyer C, Samama CM, Molliex S. Do antifibrinolytics reduce allogeneic blood transfusion in orthopedic surgery? Anesthesiology. 2006 Nov;105(5):1034-46. doi: 10.1097/00000542-200611000-00026. PMID 17065899
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Desai MH, Herndon DN, Broemeling L, Barrow RE, Nichols RJ Jr, Rutan RL. Early burn wound excision significantly reduces blood loss. Ann Surg. 1990 Jun;211(6):753-9; discussion 759-62. doi: 10.1097/00000658-199006000-00015. PMID 2357138
- [Background] Curinga G, Jain A, Feldman M, Prosciak M, Phillips B, Milner S. Red blood cell transfusion following burn. Burns. 2011 Aug;37(5):742-52. doi: 10.1016/j.burns.2011.01.016. Epub 2011 Mar 1. PMID 21367529